CLINICAL TRIAL: NCT05815017
Title: YOOMI: Effect of Gamified Physical Therapy Exercise Software on Inpatient Mobility
Acronym: YOOMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Jay Naik MD, Assistant Professor of Medicine, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro2022002225
Record Dates: First submitted 2023-03-08; First posted 2023-04-18 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Weakness, Muscle; Delirium in Old Age; Muscle Atrophy or Weakness; Muscle Loss; Hospital Acquired Condition; Physical Disability; Physical Inactivity
Keywords: Artificial Intelligence (AI); Physical Therapy; Hospitalization related muscle atrophy; Hospitalization associated decline; Inpatient rehabilitation; AI driven physical therapy
MeSH Terms: conditions — Muscle Weakness; Muscular Atrophy; Asthenia; Iatrogenic Disease; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Gamified Physical Therapy Exercise Software Intervention + Usual Care (Experimental): Participants randomized to the intervention group will be asked each day by a volunteer whether they would like to use the gamified physical therapy exercise software while in their beds. Participants willing to exercise will have the device set up for them to participate by a volunteer and the software will begin with a tutorial video for different exercises and then ask patients to perform in sequence with prompting and motion tracking. Exercises include Frontal Bicep Curls, Arm Crosses, Press Ups, Arm Rotations, and Basketball Shots.
  Interventions: Device: Yoomi Physical Therapy Software
- Usual Care (No Intervention): Usual Care

INTERVENTIONS:
Device: Yoomi Physical Therapy Software — Physical Therapy software via a computer/monitor will be set up for the patient. It will begin with a tutorial video for different exercises in the form of games and then ask patients to perform in sequence with prompting and motion tracking. Exercises include Frontal Bicep Curls, Arm Crosses, Press Ups, Arm Rotations, and Basketball Shots.
  Arms: Gamified Physical Therapy Exercise Software Intervention + Usual Care

SUMMARY:
Patients admitted to the hospital often develop functional impairments due to being in bed most of the day. Each day of bedrest leads to significant muscle loss. As a result, many patients become dependent on others or require rehabilitation at a facility to improve mobility and function prior to returning home. Staff in the hospital is limited and often unable to mobilize patients every day while hospitalized. The investigators are testing a new experimental gamified physical therapy exercise software to see if it can be a fun, enjoyable way to help mobilize patients without the assistance of staff. The primary aim of this pilot/proof of concept study is to determine whether gamified physical therapy software can help inpatients exercise within the safety of their own beds and preserve pre-hospitalization function.

ELIGIBILITY:
Inclusion Criteria:

* >= 65 years of age
* English-fluency in reading and speaking
* Capacity to consent
* Enrolled in HELP program
* Attending physician confirms there are no medical contraindications to in-bed exercises

Exclusion Criteria:

* Unstable Psychiatric Illness
* Unstable/Critically Ill Patients requiring ICU-level of care
* Surgical tube present (e.g. JP drains)
* Surgery during the hospitalization
* Bed Rest Activity Order

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction Score for Intervention Group Questionnaire (change is being assessed) | Collected daily throughout duration of patient hospitalization, usually 1-2 weeks
Software Utilization Time for Intervention Group (change is being assessed) | Collected daily throughout duration of patient hospitalization, usually 1-2 weeks
Percentage of exercise repetitions completed for Intervention Group (change is being assessed) | Collected daily throughout duration of patient hospitalization, usually 1-2 weeks
  Completed exercises divided by assigned exercises by software

SECONDARY OUTCOMES:
Patient Self-Assessments | Collected daily throughout duration of patient hospitalization, usually 1-2 weeks
  Activity Measure for Post Acute Care (AMPAC) scores done as self-assessments (Score ranging from 0 to 24 with higher being better)
3DCAM Delirium Scale | Collected daily throughout duration of patient hospitalization, usually 1-2 weeks
  22 questions including self reported and observations by staff to determine if patient has delirium
Change in Activity Measure for Post Acute Care (AMPAC) Scores | Collected daily throughout duration of patient hospitalization, usually 1-2 weeks
  Activity Measure for Post Acute Care (AMPAC) scores done by nurses twice daily (Score ranging from 0 to 24 with higher being better)
Length of hospital stay | Collected at the time of discharge of patient hospitalization, usually 1-2 weeks
Post-discharge care needs | Collected at time of discharge, usually 1-2 weeks
  Number of Partipants with Post-discharge needs e.g. subacute rehab, home PT, home assistance, acute rehab, etc
Post-discharge Self Assessed Activity Measure for Post Acute Care (AMPAC) Score | 30 days post-discharge
  AMPAC scores done as self-assessments (Score ranging from 0 to 24 with higher being better)

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Wood Johnson University Hospital, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No